CLINICAL TRIAL: NCT07375329
Title: Exploring the Utility of Breath Hydrogen and Methane as Biomarkers of Total Dietary Fiber Intake: A Pilot Study
Brief Title: Breath Hydrogen and Methane as Biomarkers of Fiber Intake
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18961
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breath Tester (Other): All participants will receive a breath tester
  Interventions: Other: Breath Tester

INTERVENTIONS:
Other: Breath Tester — Participants enrolled in a fiber-focused study will be offered a Food Marble to see if the data provided correlates with self-reported fiber intake

SUMMARY:
This study is designed to examine if mobile phone-based breath hydrogen and methane monitors can be used as a biomarker of dietary fiber intake.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in parent trial (NCT07219706)

Exclusion Criteria:

* Not enrolled in parent trial (NCT07219706)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Breath methane | Measured daily for three months
  Measured daily for three months, represented in parts per million (ppm)
Breath hydrogen | Daily for three months
  Measured daily for three months, represented in parts per million (ppm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No